ID: UMCC 2018.085 Radiotherapy, Carboplatin/Paclitaxel and Nivolumab for High Risk NCT03829722 HPV-related Head and Neck Cancer

# UNIVERSITY OF MICHIGAN CONSENT TO BE PART OF A RESEARCH STUDY

#### 1. KEY INFORMATION ABOUT THE RESEARCHERS AND THIS STUDY

#### Study title:

PHASE II TRIAL OF RADIOTHERAPY, CARBOPLATIN/PACLITAXEL AND NIVOLUMAB FOR HIGH RISK HPV-RELATED OROPHARYNX CANCER (UMCC 2018.085)

## Company or agency sponsoring the study:

The University of Michigan

#### **External support:**

Bristol Myers Squibb (BMS)

## Name, degrees, and affiliations of the principal investigator:

Michelle Mierzwa, MD

Department of Radiation Oncology, University of Michigan

## 1.1 Key Study Information

You may be eligible to take part in a research study. This form contains important information that will help you decide whether to join the study. Take the time to carefully review this information. You should talk to the researchers about the study and ask them any questions you have. You may also wish to talk to others such as your family, friends, or other doctors about joining this study. If you decide to join the study, you will be asked to sign this form before you can start study-related activities. Before you do, be sure you understand what the research study is about.

A research study is different from the regular medical care you receive from your doctor. Research studies hope to make discoveries and learn new information about diseases and how to treat them. You should consider the reasons why you might want to join a research study or why it is not the best decision for you at this time.

Research studies do not always offer the possibility of treating your disease or condition. Research studies also have different kinds of risks and risk levels, depending on the type of the study. You may also need to think about other requirements for being in the study. For example, some studies require you to travel to scheduled visits at the study site in Ann Arbor or elsewhere. This may require you to arrange travel, change work schedules, find child care, or make other plans. In your decision to participate in this study, consider all of these matters carefully.

This research is studying the addition of nivolumab to the standard of care combination of concurrent chemotherapy and radiation in small numbers of people to learn about its safety and its effect on your body at certain doses as a treatment for high risk HPV-related squamous cell carcinoma of the oropharynx (OPSCC). Nivolumab will be administered intravenously (via IV). The main purpose of this study is to see if the addition of nivolumab to the standard of care concurrent combination can improve 2-year progression free survival for high risk HPV-related OPSCC. Your health-related information and biospecimens (blood, urine, tumor tissue) will be collected for this research study.

IRBMED Informed Consent Template—3-9-2018

Instructions revised 3-9-2018

DO NOT CHANGE THIS FIELD—IRB USE ONLY

There can be risks associated with joining any research study. The type of risk may impact whether you decide to join the study. For this study, some of these risks may include serious health complications that may be life threatening, requiring hospitalization or prolonging hospitalization, no improvement of your cancer, or new symptoms from the use of the study intervention drug. More detailed information will be provided later in this document.

This study may or may not offer some benefit to you now. More information will be provided later in this document.

We expect the amount of time you will participate in the study will be 21 weeks of study intervention with follow-up visits for 2 more years.

You can decide not to be in this study. Alternatives to joining this study include standard of care therapy, radiation therapy with concurrent cisplatin, participating in another study, or palliative care.

Even if you decide to join the study now, you are free to leave at any time if you change your mind.

More information about this study continues in Section 2 of this document.

#### 2. PURPOSE OF THIS STUDY

## 2.1 Study purpose:

This is a Phase II study, which means the goal is to test the safety and effectiveness of the investigational study intervention, in other words - does it work against your type of cancer, and do the benefits outweigh the risks and side effects. This is usually done by comparing the outcomes of subjects in the study to those of people who previously received standard treatment.

The purpose of this study is to find out if the addition of nivolumab can improve 2 year progression free survival (PFS) as compared to standard of care of fractionated radiation therapy (RT) and carboplatin/paclitaxel in subjects with high risk HPV-related squamous cell carcinoma of the oropharynx (OPSCC). This standard of care combination of concurrent chemotherapy and radiation (chemoradiation) is a potentially curative therapy for oropharynx (tonsil, base of tongue, oropharyngeal wall, soft palate) cancer. Nivolumab and similar drugs have been shown to be effective in more advanced forms of head and neck cancer. Nivolumab has also been shown to be safe in addition to radiation and chemotherapy. Fractionated means the radiation will be administered in fragments or parts across multiple days. The addition of nivolumab to concurrent chemoradiation may lead to increased toxicity and a potential for dosing delays or less than optimal dosing of chemotherapy and radiation with no additional benefit compared to chemoradiation alone. None of the study drugs in combination are FDA approved for oropharynx cancer.

#### 3. WHO MAY PARTICIPATE IN THE STUDY

Taking part in this study is completely **voluntary**. You do not have to participate if you don't want to. You may also leave the study at any time. If you leave the study before it is finished, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled.

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

## 3.1 Who can take part in this study?

Subjects with squamous cell carcinoma of the oropharynx (tonsil, base of tongue, oropharyngeal wall, soft palate) that is either p16 positive or HPV positive are able to participate in this study.

Every study has strict guidelines for determining which people may participate. These are called eligibility criteria. You will need to meet all of these criteria before you can participate in this study. If you agree to consider participating in this study, you will undergo evaluations to see if you meet the eligibility criteria for this study. Even though you may meet all the criteria for participation, it is possible that you may not be enrolled in this study for other reasons.

## 3.2 How many people are expected to take part in this study?

About 40 people are expected to participate in this study, all at the University of Michigan.

## 4. INFORMATION ABOUT STUDY PARTICIPATION

## 4.1 What will happen to me in this study?

The study team will explain the research study and answer any questions you have about the study. If you still want to participate in the study the study team will request you sign the consent form prior to any activities occurring that pertain to the study. Once your consent is obtained, the study team will look through your medical chart, ask you questions, and begin scheduling tests and procedures to determine if you are eligible for the study. The study team will inform you of the types of tests and procedures required before the study begins.

Once it is determined you are eligible to enter the study, tests and procedures done at your study visits as part of your regular cancer care will continue, but some may be done more often because you are participating in this research study. Also, some of the tests or procedures may have to be repeated if, for example, they were done too long ago or the results are not normal.

Some tests and procedures may be done that are not part of your regular cancer care and are being done only for this research study. Tests and procedures that are performed more often or are not part of your standard cancer care will be identified below as "Research".

#### During the study you must:

- Follow the instructions you are given.
- Come to the study center for your visits with the study doctor.
- Tell the study doctor or study staff about any changes in your health and/or medications you are taking.
- Tell the study doctor or study staff if you want to stop being in the study at any time.

#### Before starting the study

You will need to have the following exams, tests or procedures to find out if you can be in this study and before beginning study intervention. If you have had some of them recently, they may not need to be repeated. The screening tests and procedures do not have to be completed in one day and you are allowed to take breaks if you have multiple procedures in one day.

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

Before you begin the study you will need to have the following screening procedures:

- Medical history: including any past treatments, surgeries, infection, autoimmune diseases and smoking history.
- Medications: It is important that you tell your doctor about all of the medications that you have been taking, including over the counter medicines, vitamins or herbal treatments.
- Physical exam: including measurement of your height, weight, blood pressure, heart rate, respiratory rate and temperature.
- Performance status: Your ability to perform day to day activities and care for yourself
- Routine blood tests (approximately 2 teaspoons): will be drawn for tests to check blood counts and chemistry
- **OPTIONAL blood test:** see Samples Stored for Genetic Testing below (RESEARCH)
- Scans of your cancer:
  - Magnetic Resonance Imaging (MRI) scan takes an image of your head or body to observe the location and size of your tumor. For the MRI scan, you may be given a "contrast material" (a special dye that makes it easier for doctors to see different tissues in your body). You will be asked to lie down on a narrow bed which will slide into a tunnel that is 6 feet long by 22 inches across and is open at each end. You will be asked to lie quietly for about one hour, during which time you will hear a loud machinelike noise. A MRI scan takes about an hour and a half to complete. (RESEARCH)
  - PET/CT scan makes detailed, computerized pictures that helps reveal how your tissues are functioning. For at least 4 hours before the PET/CT scan, you must not eat or drink anything except water. A small tube will be placed in your arm, and you will receive an injection of a very small amount of a mildly radioactive material into your bloodstream. The radioactive nature of this injected material allows the scanner to "see" it in certain places in your body. After the injection, you will need to rest quietly until it is time for the scan. The amount of rest time may vary, but be prepared to wait for between 45 and 90 minutes. During the scan, you will lie flat on your back on a table. The scan itself may last up to 1 hour. (some of these are for RESEARCH)
- **Videofluoroscopy**: to evaluate swallowing problems from radiotherapy, you will undergo an evaluation of swallowing by videofluoroscopy (VF). VF consists of swallowing a small quantity of barium, or a barium-coated food such as a cookie, while a series of x-rays are taken of the throat.
- **Urine pregnancy test for Women of Child Bearing Potential**
- **Dental exam**
- Quality of life (QOL) questionnaire (RESEARCH)
- **Nutritional assessment**
- **Tumor specimen:** Your study doctor will request original tumor samples (called archival tissue) from a previous biopsy. By signing this consent, you provide your permission to obtain these original samples and allow your study doctor to submit them for sequencing analysis. If you do not have archival tissue available, you will be asked to undergo a fresh tissue biopsy.

Some of the above procedures will be performed at additional time points during your participation in this study. Please see the table on the following page for more information.

Instructions revised 3-9-2018 DO NOT CHANGE THIS FIELD-IRB USE ONLY

#### **Study Intervention**

You will start study intervention within 30 days of enrollment. On Day 1 you will receive nivolumab 240 mg intravenously (via IV, meaning it's given through a vein in your arm), and then continuing every 2 weeks throughout Radiation Therapy for 4 doses. No radiation will be given on Day 1.

On day 8 you will receive paclitaxel (30mg/m²) via IV, followed directly by carboplatin (AUC=1) via IV, and then a 1-hour observation period. You will then receive Radiation Therapy (70 gray in 35 daily fractions on business days, Monday-Friday) beginning within 24 hours of carboplatin/paclitaxel administration. Carboplatin/paclitaxel will be administered weekly during Radiation Therapy. On days you receive nivolumab it will be given before carboplatin/paclitaxel administration. You will receive a total of 7 concurrent carboplatin/paclitaxel and 4 concurrent nivolumab doses. Starting in week 9, after completing Radiation Therapy, you will receive nivolumab (480 mg) every 4 weeks for a total of 4 doses.

 Consent Subtitle: UMCC 2018.085 Consent Version: ICF v18Sep2020

## The table below describes the procedures that will be completed at each of the visits.

| | Screen<br>ing | Pre-<br>Thera<br>py | Day 1 | Pre-RT | Between fractions 8-12 | Weekly<br>during<br>CRT* | + 1<br>Month <sup>1</sup> | + 3<br>month <sup>1</sup> | + 6<br>month <sup>1</sup> | + 12<br>month <sup>1</sup> | + 24<br>month <sup>1</sup> | Recurrence<br>** |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Rad Onc evaluation | Х | Х | | | | Χ | Х | Х | Х | Х | Χ | X |
| CBC with diff, CMP, | | | | | | | | | | | | |
| Mg, LFTs, TSH, | Х | Х | | | | $\chi_3$ | X3 | X3 | X | Х | | |
| cortisol <sup>2</sup> | | | | | | | | | | | | |
| Pregnancy test <sup>4</sup> | Х | | | | | | | | | | | |
| MRI (R) | | <b>X</b> <sup>5</sup> | | | <b>X</b> <sup>5</sup> | | | | | | | |
| PET/CT | Х | Х | | | X (R) | | | Х | | | | Х |
| Toxicity & nutritional | | V | | V | | V | V | | V | V | V | |
| Evaluation | | X | | Х | | X | Х | Х | Х | X | Х | |
| Quality of Life | | Х | | Х | | Х | х | х | х | Х | | |
| Questionnaire <sup>6</sup> (R) | | _ ^ | | ^ | | ^ | ^ | ^ | _ ^ | ^ | | |
| Videofluoroscopy | | Х | | | | | | Х | | Х | | |
| Dental | | | | Х | | | | | | | | |
| Evaluation <sup>7</sup> | | | | ^ | | | | | | | | |
| Carboplatin/paclitaxel | | | | | | Χ | | | | | | |
| Nivolumab | | | Х | | | X <sub>8</sub> | X <sup>9</sup> | | | | | |
| OPTIONAL: Blood | | V | | | | V | V | | V | V | V | V |
| correlative studies (R) | | Х | | | | Х | X | X | X | X | Х | Х |
| Primary tumor | | | | | | | | | | | | |
| specimen for | | X <sup>10</sup> | | | | | | | | | | X <sup>10</sup> |
| correlatives required | | | | | | | | | | | | |

- 1 Radiation oncology (RadOnc) exam will include medical history and physical as well as pregnancy test if applicable. RadOnc evaluation must be completed at baseline and will include smoking history. Follow-up visits may be completed by RadOnc, Otolaryngology, or Medical Oncology.
- 2 Baseline within 2 weeks of registration
- 3 Labs during RT, and in follow up 1-mo through 3-mo will occur with each chemotherapy dose
- 4 Pregnancy test should also be performed as part of pre-RT workup in women of child bearing potential
- 5 MRI is encouraged but not required- patients with a contraindication to MRI or who are unable to tolerate MRI will continue on the study as otherwise planned
- 6 QOL suggested but not required.
- 7 Pre-RT dental evaluation is encouraged but not required.
- 8 Nivolumab will be started on Day 1 and given every 2 weeks for 4 total doses concurrent with RT.
- 9 Following completion of RT, nivolumab will be given every 4weeks for a total of 4 doses.
- 10 Biopsy is strongly encouraged; archival tissue is acceptable
- \* CRT=chemoradiation
- \*\* Recurrence is cancer found afterstudy intervention, and after a period of time when the cancer couldn't be detected.
- (R) RESEARCH

## **Follow-Up and Recurrence**

You will return to the clinic for follow-up visits 3, 6, 12, and 24 months following completion of Radiation Therapy. If your cancer recurs after study intervention you will return to the clinic. Refer to the table above for Follow-Up and Recurrence procedures that will be performed.

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

## **OPTIONAL: Blood Samples Stored for Genetic Testing (RESEARCH)**

Blood samples will be collected at routine time points during the course of this study as described above. These samples and related medical information (for example, your diagnosis, disease history, prior treatment, etc.) will be stored for future research testing. The purpose of the research testing on your blood samples is to study how your genes affect the way your cancer responds to the study intervention. Researchers want to see if recurrent cancer in HPV positive OPSCC can be detected in blood and if it can identify tumor recurrence earlier than clinical exam. You can take part in this study even if you decide not to let us analyze your blood to find out if recurrent cancer in HPV positive OPSCC can be detected in blood and if it can identify tumor recurrence earlier than clinical exam.

About 6 ½ teaspoons of blood will be collected at screening, weekly during study intervention, and at 4 weeks, 3 months, 6 months, and 12 months post-therapy for genetic testing. About 78 teaspoons of blood total will be collected for genetic testing.

For comparison, the standard blood donation is about 2 cups collected at once.

Your samples will be kept at the Brenner/Walline/Zhou labs at the University of Michigan. The University of Michigan will control the samples, and they will be stored indefinitely or until they are used up.

Even if you give us permission now to keep some of your samples and related medical information, you can change your mind later and ask us to destroy it. Keep in mind, however, that once we have analyzed your samples, we may not be able to take the information out of our research. Also, if we have shared some of your samples and related medical information with other researchers, we will not be able to get it back.

For blood draw risks please refer to Section 5.1 of this consent form. For information related to loss of confidentiality and genetic risks, please refer to Section 9.1 of this consent form.

We will not tell you the results of the future analysis of your blood samples. Allowing us to do future research on your blood samples and related medical information will not benefit you directly.

The University of Michigan or the investigators or study team may benefit financially from future research on your blood samples and related medical information.

As part of this study, your coded results may be shared with BMS.

With appropriate permissions, your coded samples and collected information may also be shared with other researchers, here, around the world, and with companies.

Your identifiable private information or identifiable biospecimens may be stripped of identifiers and used for future research studies or distributed to another researcher for future research studies without additional informed consent.

IRBMED Informed Consent Template—3-9-2018

Instructions revised 3-9-2018

DO NOT CHANGE THIS FIELD—IRB USE ONLY

Research can lead to new discoveries, such as new tests, drugs, or devices. Researchers, their organizations, and other entities, including companies, may potentially benefit from the use of the data or discoveries. You will not have rights to these discoveries or any proceeds from them.

You can make your choice in Section 12 of this form.

## **Tumor Tissue for Unspecified Future Research (RESEARCH)**

Besides the information about the main study, the following information is specific to unspecified future use of identifiable data and/or biospecimens. We will keep some of your tumor tissue and medical information collected in the main study, so that we may study it in future research. The future research may be similar to this study or may be completely different.

We will use your tumor tissue and medical information for future research. Even if you give us permission now to keep some of your tumor tissue and medical information, you can change your mind later and ask us to destroy it. Keep in mind, however, that once we have analyzed your tumor tissue, we may not be able to take the information out of our research.

We may share your tumor tissue and medical information with other researchers, so that they can use it in their research. Their research may be similar to this study or may be completely different. Once we have shared your tumor tissue and medical information with other researchers, we will not be able to get it back.

For information related to loss of confidentiality and genetic risks, please refer to Section 9.1 of this consent form. Future use of your identifiable data and/or specimens will be conducted in compliance with applicable regulatory requirements.

Instructions revised 3-9-2018

DO NOT CHANGE THIS FIELD—IRB USE ONLY

You will not find out the results of future research on your tumor tissue. Allowing us to do future research on your tumor tissue and medical information will not benefit you directly.

With appropriate permissions, your samples and collected information may also be shared with other researchers here, around the world, and with companies.

Your identifiable private information or identifiable biospecimens may be stripped of identifiers and used for future research studies or distributed to another researcher for future research studies without additional informed consent.

Research can lead to new discoveries, such as new tests, drugs, or devices. Researchers, their organizations, and other entities, including companies, may potentially benefit from the use of the data or discoveries. You will not have rights to these discoveries or any proceeds from them.

You will be asked to affirm in Section 12 of this consent form your required permission to keep your tumor tissue and related medical information for future research.

## 4.2 How much of my time will be needed to take part in this study?

Screening and pre-therapy activities may take about 5-7 hours and do not need to be completed in one day.

Your Day 1 clinic visit may take about 4-5 hours.

Pre- radiation therapy activities may take about 2-3 hours. These procedures are standard of care.

Your MRI and PET/CT visit between fractions 8-12 may take about 3-5 hours. These studies are for research only.

Weekly clinic visits during radiation therapy for carboplatin/paclitaxel infusions may take about 5-7 hours. Clinic visits during radiation therapy beginning with nivolumab infusions followed by carboplatin/paclitaxel infusions may take about 6-8 hours.

Follow-up visits at 3, 6, 12, and 24 months following completion of Radiation Therapy may take about 3-4 hours. The +3 Month visit may take about 7-8 hours in order to complete a PET scan, clinic visit with physician, blood collection and swallow study (these are standard) as well as quality of life surveys for the study.

A clinic visit at recurrence may take about 5-6 hours.

## 4.3 When will my participation in the study be over?

Study intervention will continue for 21 weeks total, and follow-up visits will continue up to 2 more years.

#### 4.4 What will happen with my information and/or biospecimens used in this study?

Your biospecimens and collected information may be shared with BMS.

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

With appropriate permissions, your biospecimens and collected information may also be shared with other researchers, here, around the world, and with companies.

Your identifiable private information or identifiable biospecimens may be stripped of identifiers and used for future research studies or distributed to another researcher for future research studies without additional informed consent.

## 5. INFORMATION ABOUT STUDY RISKS AND BENEFITS

## 5.1 What risks will I face by taking part in the study? What will the researchers do to protect me against these risks?

The known or expected risks are:

#### Risks and Side Effects Related to Radiation Therapy of the Oropharynx

## Very Likely (≥10 of subjects)

- Sores in the mouth and/or throat which can be painful and make it very difficult to chew and or swallow foods
- Mouth dryness or changes in taste and/or smell that may be permanent
- Thick saliva
- Hoarseness
- Tanning or redness and/or irritation of the skin in the head and neck area being treated with radiation
- Ear pain and/or pressure
- Fatigue
- Weight loss
- Permanent hair loss in the area treated with radiation (face, chin, neck)
- Loss of teeth, or cavities in the teeth, if strict dental care is not followed and/or hypersensitivity
  of teeth

## Less Likely, But Serious (1-9% of subject; except if noted)

- Decrease in function of the thyroid gland that may require you to take thyroid replacement medicine to prevent you from feeling tired or sleepy
- Serious damage to the nerves in the neck, jawbone, voice box, skin, or other parts of the head and neck that may require a major operation to correct and, rarely, can even be life threatening (1-5% of subjects)
- Temporary pain or scarring around nerves in the shoulder that could cause numbness and/or weakness
- Breathing problems
- Difficulty with swallowing and eating for which you might need a long term or permanent feeding tube; possibility of inhaling food and/or liquids into the lungs – which could also result in pneumonia.
- Serious ear infections and/or hearing loss
- Damage to the spinal cord leading to permanent weakness and/or symptoms like a "stroke". This is a very rare complication occurring in < 1% of patients.

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

• Stroke has been reported to be slightly higher after head and neck radiation, compared with the general population, due to the possibility of increased formation of plaque in the carotid artery (causing blockage). Your doctors will monitor for carotid blockage with ultrasound.

## **Risks and Side Effects Related to Carboplatin**

## **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Carboplatin, more than 20 and up to 100 may have:

- Hair loss
- Vomiting, nausea
- Infection, especially when white blood cell count is low
- Anemia which may cause tiredness, or may require blood transfusions
- · Bruising, bleeding
- Belly pain

## **OCCASIONAL, SOME MAY BE SERIOUS**

In 100 people receiving Carboplatin, from 4 to 20 may have:

- Diarrhea, Constipation
- Numbness and tingling in fingers and toes
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Changes in taste
- Changes in vision

## **RARE, AND SERIOUS**

In 100 people receiving Carboplatin, 3 or fewer may have:

• Damage to organs which may cause hearing and balance problems

## **Risks and Side Effects Related to Paclitaxel**

## **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Paclitaxel, more than 20 and up to 100 may have:

- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Infection, especially when white blood cell count is low
- Bruising, bleeding
- Anemia which may cause tiredness, or may require blood transfusions
- Pair
- · Sores in mouth which may cause difficulty swallowing
- Diarrhea, nausea, vomiting
- Muscle weakness
- Numbness, tingling or pain of the arms and legs
- Hair loss

IRBMED Informed Consent Template — 3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD — IRB USE ONLY

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving Paclitaxel, from 4 to 20 may have:

- Abnormal heartbeat
- Blood clot which may cause swelling, pain, shortness of breath
- Damage to the lungs which may cause shortness of breath

#### RARE, AND SERIOUS

In 100 people receiving Paclitaxel, 3 or fewer may have:

- Heart attack or heart failure which may cause shortness of breath, swelling of ankles, and tiredness
- A tear or a hole in the bowels which may cause pain or that may require surgery
- Severe skin rash with blisters and peeling which can involve mouth and other parts of the body

#### **Risks and Side Effects Related to Nivolumab**

#### **Risks of Nivolumab**

Nivolumab may cause one or more of the side effects listed below. This information is based on data from cancer subjects in clinical trials with nivolumab. In addition, there may be side effects that are not yet known that may occur. You should tell your doctor or nurse right away about any possible side effects you experience.

Very common (≥10% of subjects)

- Diarrhea
- Feeling tired or lack of energy
- Skin itching
- Skin rash

## Common side (≥1% to <10% of subjects)

- Abdominal pain
- Alkaline phosphatase increased: lab test result associated with liver or bone abnormalities
- Allergic reaction/hypersensitivity
- ALT increased: lab test result associated with abnormal liver function
- Amylase increased: lab test result associated with pancreas inflammation
- AST increased: lab test result associated with abnormal liver function
- Bilirubin increased lab test result associated with abnormal liver function
- Chills
- Constipation
- Cough
- Creatinine increased: lab test result associated with decreased kidney function
- Decreased appetite
- Dizziness or vertigo (feeling off balance which can lead to dizziness)
- Dry mouth
- Dry skin
- Fever

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

 Consent Subtitle: UMCC 2018.085
Consent Version: ICF v18Sep2020

- Headache
- Increased blood sugar
- Inflammation of the colon (colitis)
- Inflammation of the mouth
- Infusion related reaction
- Lipase increased: lab test result associated with pancreas inflammation
- Loss of color (pigment) from areas of skin
- Low levels of sodium in the blood
- Low platelet counts (thrombocytopenia): this may increase your risk for skin bruising, nose bleeds, and bleeding from the gums
- Low red blood cell counts (anemia): this may make you feel weak and tired
- Lung inflammation (pneumonitis): it is possible that nivolumab may cause inflammation of the
  tissues of the lung. This adverse effect has been reported in patients treated with nivolumab.
  While many patients with X-ray or CT abnormalities have not developed any symptoms, some
  patients have developed mild to severe symptoms and in rare cases, death has occurred as a
  result of their lung inflammation. Signs and symptoms of lung inflammation may include
  difficulty breathing, pain or discomfort while breathing, chest pain, cough, shortness of breath,
  increased rate of breathing, fever, low blood oxygen levels, or fatigue
- Nausea
- Pain in the muscles, bones, ligaments, tendons, and nerves
- Reaction related to infusion of the medicine. The symptoms may include but not limited to fever, rash, pain, swelling
- Redness of the skin
- Renal (kidney) failure or damage to your kidneys
- Shortness of breath
- Sodium levels in the blood low
- Swelling, including face, arms, and legs (oedema)
- Thyroid gland function decreased or may be increased; increased thyroid stimulating hormone-a lab test results associated with abnormal thyroid function
- Thyroid stimulating hormone increased: lab test result associated with abnormal thyroid function
- Tingling, burning, numbness or weakness, possibly in arms, legs, hands and feet
- Vomiting

#### Uncommon (≥0.1% to <1% of subjects)

- Bronchitis: inflammation of the lining of bronchial tubes, which carry air to and from the lungs
- Decreased secretion of hormones produced by adrenal glands
- Decreased thyroid stimulating hormone a lab test result associated with abnormal thyroid function
- Dehydration
- Diabetes: a disease that results in too much sugar in the blood
- Dry eyes
- Erythema multiforme: a skin disorder that is considered to be an allergic reaction to medicine
  or an infection. Symptoms may include symmetrical, red raised skins areas that can appear
  all over the body, more noticeable on the fingers and toes. These patches often look like

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

"targets" (dark circles with purple-grey centers)

- Heart rate increased
- Heart rhythm abnormal
- High blood pressure
- Hives
- Inflammation of the eye
- Inflammation of the kidney
- Inflammation opituif the pancreas
- Inflammation of the pituitary gland
- Inflammation of the stomach
- Inflammation of the thyroid gland
- Joint pain or stiffness
- Kidney function failure, kidney disease
- Liver inflammation
- Low blood pressure
- Low white blood cell counts (neutropenia): these put you at higher risk for infection
- Pemphigoid: blistering of the skin or mouth caused by the immune system attacking healthy tissue
- Respiratory failure: a condition in which not enough oxygen passes from your lungs into your blood, or when your lungs cannot properly remove carbon dioxide
- Skin disease with thickened patches of red skin, often silvery scales (Psoriasis)
- Trouble falling and/or staying asleep (Insomnia)
- Underactive function of the pituitary gland situated at the base of the brain
- Upper respiratory tract infection: A common viral / bacterial infection that affects the nose, throat, and airways
- Vision blurred

## Rare (≥0.01% to <0.1% of subjects)

- Autoimmune hemolytic anemia: a malfunction of the immune system that produces autoantibodies, which attack red blood cells as if they were foreign substances to the body
- Cranial nerve disorder
- Damage to the protective covering of the nerves in the brain and spinal cord
- Diabetes complications resulting in excess blood acids and diabetic coma
- Disease caused by the body's immune system attacking healthy organs
- Double vision
- Drug induced liver injury
- Guillain-Barre syndrome, an autoimmune disorder associated with progressive muscle weakness or paralysis
- Histiocytic necrotizing lymphadenitis or Kikuchi lymphadenitis: disorder of the lymph nodes
  which causes the lymph nodes to become enlarged, inflamed and painful, commonly affecting
  nodes of the neck and possibly associated with fever or muscle and joint pains
- Inflammation of blood vessels
- Inflammation of the heart
- Inflammation of the lining of the brain and spinal cord
- Lung infiltrates, associated with infection or inflammation

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

- Muscle inflammation
- Myasthenic syndrome (neurologic syndrome characterized by muscle weakness) including myasthenia gravis, a nerve disease that may cause weakness of eye, face, breathing, and swallowing muscles.
- Pericarditis: a swelling and irritation of the thin saclike membrane surrounding the heart (pericardium)
- Polymyalgia rheumatica, an inflammatory disorder causing muscle pain and stiffness
- Rhabdomyolysis: muscle fiber released into the blood stream which could damage your kidneys
- Rosacea: acne-like skin condition resulting in redness of face
- Rupture of the intestine/hole in the intestine
- Sarcoidosis, a disease involving abnormal collections of inflammatory cells (granulomas) in organs such as lungs, skin, and lymph nodes
- Severe allergic reaction may include but not limited to high grade fever, rash, swelling and pain
- Stevens Johnson syndrome: inflammatory disorder of skin and mucous membranes, resulting in blistering and shedding of skin
- Toxic epidermal necrolysis: a potentially fatal disease characterized by blistering and peeling of the top layer of skin resembling a severe burn

The following events have been identified during post-approval use of nivolumab. Because reports are voluntary from a population of unknown size, an estimate of frequency cannot be made.

- Graft-versus-host-disease: a condition that occurs when donor bone marrow or stem cells attack the recipient.
- Hemophagocytic lymphohistiocytosis (HLH) syndrome: a disease that may affect your body's
  defense system, called the immune system. Certain white blood cells may attach other blood
  cells. These abnormal blood cells collect in your spleen and liver, causing these organs to
  enlarge. The symptoms may include fever, rash, and low blood cell counts.
- Solid organ transplant rejection
- Vogt-Koyanagi-Harada (VKH) disease: a disease that may affect several parts of the body, including the eyes, ears, nervous system, and skin. The symptoms may include eye swelling, pain and/or blurred vision; hearing loss, ringing in the ears; and /or loss of skin color.

## Additional information on pneumonitis:

Your study doctor and nurse will watch you closely for changes in your ability to breathe and for other signs or symptoms that might show you are developing this type of lung inflammation and will perform regular tests including physical exams, measurement of oxygen levels through non-invasive testing (i.e., pulse oximeter), blood tests, chest x-rays and/or CT scans.

## Please inform your study doctor or nurse AT ONCE if you experience any of the following:

- Any new or increased shortness of breath;
- Any new or increased chest pain;
- Any new or increased pain/difficulty while breathing;
- Any new or increased cough or any significant change in your type of cough; for example, any new or increased mucous or blood in your cough;

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

 Consent Subtitle: UMCC 2018.085
Consent Version: ICF v18Sep2020

- Any change in the amount of oxygen you require;
- Any fever, fatigue, or other symptoms that occur at the same time as any changes to your breathing or other lung symptoms.

If you start to develop symptoms, your study doctor will ask you to return to the clinic for additional tests, which could include a physical exam, measurement of oxygen levels, blood tests, chest x-rays, and/or CT scans. You will be monitored very closely for changes in your overall lung symptoms, monitoring may require hospitalization. You may require specific treatment in order to control pneumonitis. You may also be seen by a special doctor called a pulmonologist, who has special training to be an expert in how your lungs work.

Prolonged treatment with medicines that suppress inflammation, sometimes needed to manage the side effects of nivolumab study intervention, may lower your body's ability to fight off certain infections (i.e., opportunistic infections). These infections may require treatment with antibiotic or antifungal medications and may be fatal.

Complications, including fatal events, have occurred in patients who received allogeneic hematopoietic stem cell transplantation (HSCT) after nivolumab.

Complications, including rejection, have also been reported in patients who have received an organ or tissue transplant. Study intervention with nivolumab may increase the risk of rejection of the organ or tissue transplant.

#### **Other Side Effects**

#### **Blood Draws**

Collection of blood samples may cause pain, bleeding, bruising or infection. It is also possible that you may feel lightheaded or faint. Please tell your study doctor or the study nurse if you do not feel well after having your blood drawn at any time during your study participation.

### **Tumor Biopsy**

A piece of a tumor will be removed for testing. Potential risks and discomforts that you may experience as a result of the procedure depend upon the location of the tumor. The more common risks/discomforts include pain, bleeding, infection, damage to tissues, and healing complications. Your doctor will further explain any specific risks that may apply based on the procedure, and you will sign a separate consent for the procedure which will provide risk information in more detail. In order to make the procedure more comfortable, you will get a local anesthetic to numb the area. A mild sedative may also be given to you.

## Questionnaires

As part of the study, you will be asked to complete questionnaires. Some of the questions may seem very personal or embarrassing. They may make you uncomfortable. You may refuse to answer any of the questions that you do not wish to answer.

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

#### **MRI Risk**

MRIs done for research that use IV contrast have risks similar to MRIs done for clinical care. Contrast is used to improve the pictures of the inside of the body made by the MRI. Common risks of MRI include: feeling fearful of being in a small enclosed space (claustrophobia) when you are lying inside the MRI scanner, feeling uncomfortable because of the loud noises made by the machines, and feeling uncomfortable with the physical sensations you may feel during the process. You are also exposed to some risk because of the injected contrast, gadolinium-DTPA, which may cause headache, nausea, and local burning sensation.

The contrast agent, gadolinium has been linked to development of Nephrogenic Fibrosing Dermopathy (NFD), also known as Nephrogenic Systemic Fibrosis (NSF). NFD is a thickening of the skin, organs and other tissues and is a rare complication in subjects with kidney disease who undergo an MRI with contrast material. To help prevent this, we will check how well your kidneys work before you have any MRIs. Because of the use of contrast, all female subjects who are able to have children will be required to use adequate birth control. If you have implanted metal objects such as a pacemaker, artificial limbs, or metal joints, you will not be able to have an MRI done, and may not be able to take part in this research.

#### **PET-CT Scan**

A PET-CT (positron emission tomography-computed tomography) scan is a nuclear medicine imaging test performed with a CT scan. The combined images show the location of abnormal metabolic activity within the body. A small amount of radioactive material (radiopharmaceutical or radiotracer) is injected intravenously before imaging for the PET component of the test. Radiation emitted from the radiotracer is detected by a special camera or imaging device called a PET scanner. The radiotracer used in this study is  $2-[^{18}F]$  fluoro-2-deoxy-D-glucose ( $[^{18}F]$  FDG), a radioactive form of sugar. The CT uses ionizing radiation to obtain pictures of the body. Everyone is exposed to naturally occurring ionizing radiation every day, which is called 'background radiation'. The biological effect of radiation exposures in humans is measured in terms of Sieverts (Sv) or milliSieverts (1 mSv = 1/1000 Sv), which is a unit of uniform whole body radiation exposure. For each PET/CT scan you have with [18F]FDG, your radiation exposure will be approximately 11 mSv from internal and external exposures. The natural background radiation you are exposed to, like everyone else living on this planet, is on average 3 mSv per year. The radiation you will be exposed to for each PET/CT scan is equal to 3.7 times this yearly background radiation. The U.S. Federal Government requires that the annual amount of radiation exposure of radiation workers must not exceed 50 mSv per year; the radiation you will be exposed to from each PET/CT scan in this study is equal to 22% of this amount.

Your lifetime radiation risk also includes any radiation you may have received in the past for diagnosis or treatment, and any such radiation you may be exposed to in the future. Please inform the investigators if you have had any major radiation exposure in the past, particularly in the past year, such as medical treatment with X-rays or radioactivity, or diagnostic X-rays, CT scans, or nuclear medicine scans.

No PET studies will be performed on pregnant, nursing, or potentially pregnant women, as determined by pregnancy testing within 48 hours prior to the PET scanning session.

IRBMED Informed Consent Template—3-9-2018

Instructions revised 3-9-2018

DO NOT CHANGE THIS FIELD—IRB USE ONLY

## Videofluoroscopy

There is a slight chance of cancer from excessive exposure to radiation. Some subjects may be allergic to the flavoring added to some brands of barium. If barium accidentally gets into your lungs because you aspirate during the exam, it does not cause any lasting harm, however barium may be visible on future images. There is a slight chance that barium could be retained in your gastrointestinal (GI) system leading to a blockage. If you have a known obstruction in your GI tract you should not undergo this exam.

## **Reproductive Risks**

#### Women

If there is ANY chance that you can get pregnant, you must either agree to not have vaginal intercourse or you must use TWO types of birth control (one from each list below) AT THE SAME TIME. These birth control methods must be used from the time of enrollment, all during study intervention including during temporary breaks from therapy, and for at least 5 months after your last dose of nivolumab. The following methods are considered acceptable birth control methods:

## **Primary forms**

- tubal sterilization (tubes tied)
- partner's vasectomy
- intrauterine device

## Secondary forms

- •male latex condom with or without spermicide
- •diaphragm with spermicide
- •cervical cap with spermicide
- vaginal sponge (contains spermicide)

Any birth control method can fail. The reports of birth control failing are more frequent for female patients who use only a single form of birth control. Using two forms of birth control at the same time greatly reduces the chances of pregnancy.

Additionally, you should not breastfeed during study intervention with nivolumab and carboplatin/paclitaxel, and should not resume breastfeeding earlier than 60 days following your last dose of carboplatin/paclitaxel.

#### Men

Men must agree to either abstain from sexual activities that could result in pregnancy or use an acceptable form of birth control while taking part in the study. Acceptable forms of birth control are male latex condom (with or without spermicide) or vasectomy. Men who are receiving nivolumab and who are sexually active with women of child bearing potential will be instructed to adhere to contraception for a period of 7 months after the last dose of nivolumab.

## These risks will be minimized by:

We will minimize the risks by monitoring you carefully. We will provide the usual supportive care that would be routinely given to someone with your condition. If you have side effects from the investigational study treatment, we will make appropriate adjustments as defined by the study protocol. You may need to discontinue the investigational study treatment if the side effects are too serious. If you have signs of infection, you will receive appropriate antibiotics. If you have signs of bleeding you may need to receive transfusions of platelets, plasma, or red cells. If you start feeling sick to your

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

stomach, you may be given medications to help reduce nausea. If you have vomiting, you may be given fluids through an IV.

Additionally, there may be a risk of loss to confidentiality or privacy. See Section 9 of this document for more information on how the study team will protect your confidentiality and privacy.

As with any research study, there may be additional risks that are unknown or unexpected.

## 5.2 What happens if I get hurt, become sick, or have other problems as a result of this research?

The researchers have taken steps to minimize the risks of this study. Even so, you may still have problems or side effects, even when the researchers are careful to avoid them. Please tell the researchers listed in Section 10 about any injuries, side effects, or other problems that you have during this study. You should also tell your regular doctors.

If you think you have an injury or illness that is related to your participation in this clinical trial, it is important that you tell your study doctor immediately. If you have a clinical trial related injury or accident, the study staff will make sure that you get medical treatment.

You will receive appropriate medical care for any side affects you have while participating in this study. Your study doctor may also lower the drug dose or stop drug if you experience side effects.

You must inform your study doctor immediately if there are any changes in your health/condition, or if you have any concerns regarding the study. If for any reason you are seen by another healthcare provider or admitted to another hospital, you should make known your participation in this research study. These healthcare providers may wish to contact your study doctor to discuss your condition. Your study doctor may need to contact your other doctors if you develop any potentially significant, unexpected diseases or conditions that may have been caused by the study intervention or procedures or are discovered during the study.

#### 5.3 If I take part in this study, can I also participate in other studies?

<u>Being in more than one research study at the same time, or even at different times, may increase the risks to you. It may also affect the results of the studies</u>. You should not take part in more than one study without approval from the researchers involved in each study.

#### 5.4 How could I benefit if I take part in this study? How could others benefit?

You may not receive any personal benefits from being in this study. However, others may benefit from the knowledge gained from this study.

## 5.5 Will the researchers tell me if they learn of new information that could change my willingness to stay in this study?

Yes, the researchers will tell you if they learn of important new information that may change your willingness to stay in this study. If new information is provided to you after you have joined the study, it is possible that you may be asked to sign a new consent form that includes the new information.

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

#### 6. ALTERNATIVES TO PARTICIPATING IN THE STUDY

## 6.1 If I decide not to take part in this study, what other options do I have?

If you decide not to participate, you will be treated with the best standard therapy, according to the clinical judgment of your physicians. Other treatments available for your condition include:

- Radiation therapy with concurrent cisplatin
- Taking part in another study
- Getting comfort care, also known as palliative care. This type of care helps reduce pain, tiredness, appetite problem and other problems caused by cancer. It does not treat the cancer.

## 7. ENDING THE STUDY

## 7.1 If I want to stop participating in the study, what should I do?

You are free to leave the study at any time. If you leave the study before it is finished, there will be no penalty to you. You will not lose any benefits to which you may otherwise be entitled. If you choose to tell the researchers why you are leaving the study, your reasons for leaving may be kept as part of the study record. If you decide to leave the study before it is finished, please tell one of the persons listed in Section 10 "Contact Information".

You are free to partially or completely end your participation in the study. An example of partially ending your participation would be to discontinue receiving study intervention, while still allowing continuation of study follow-up procedures.

Please note that any information collected before you withdraw will be kept and used to complete the research.

Please note that even if you withdraw consent for further follow-up or contacts, if the study doctor becomes aware of additional safety information this will be reported to the sponsor in order to comply with legal or regulatory requirements.

## 7.2 Could there be any harm to me if I decide to leave the study before it is finished?

You are free to leave the study at any time. If you leave the study before it is finished, there will be no penalty to you. This will not affect your future medical care in any way and you will not lose any benefits to which you may otherwise be entitled. Tell the study doctor if you are thinking about stopping or decide to stop. It is important to tell the study doctor if you are thinking about stopping so any risks can be evaluated by your doctor. He or she will also tell you how to stop safely and discuss what follow-up care and testing could be most helpful for you. If you choose to tell the researchers why you are leaving the study, your reasons for leaving may be kept as part of the study record. If you decide to leave the study before it is finished, please tell your study doctor or one of the researchers listed in Section 10 "Contact Information".

## 7.3 Could the researchers take me out of the study even if I want to continue to participate?

Yes. There are many reasons why the researchers may need to end your participation in the study. Some examples are:

- The researcher believes that it is not in your best interest to stay in the study.
- You become ineligible to participate.

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

- Your condition changes and you need treatment that is not allowed while you are taking part in the study.
- You do not follow instructions from the researchers.
- The study is suspended or canceled.

### 8. FINANCIAL INFORMATION

## 8.1 Who will pay for the costs of the study? Will I or my health plan be billed for any costs of the study?

The study will pay for research-related items or services that are provided only because you are in the study. If you are not sure what these are, see Section 4.1 above or ask the researchers for a list. If you get a bill you think is wrong, call the researcher's telephone number listed in Section 10.1.

BMS will provide nivolumab at no cost to you.

You or your health plan will pay for all the things you would have paid for even if you were not in the study, like:

- Carboplatin
- Paclitaxel
- Health care given during the study as part of your regular care
- Items or services needed to give you study drugs or devices
- Monitoring for side effects or other problems
- Deductibles or co-pays for these items or services.

If you do not have a health plan, or if you think your health plan may not cover these costs during the study, please talk to the researchers listed in Section 10 below or call your health plan's medical reviewer.

The study team has given you instructions about this research study. It is important that you follow these instructions carefully. If you get sick, have a medical complication, or are injured as a result of your being in the study, call Dr. Mierzwa, at (734) 936-4300 or at (734) 936-4000 (Hospital Operator – 24-hour paging). The doctor will either treat you or send you to another doctor for treatment.

If you are injured or in the event of a medical emergency, dial 911 or visit your nearest Emergency Room. If you believe the study has made you sick or caused you injury, contact one of the people listed in section 10 of this document (Contact Information). If taking part in the study makes you sick or causes you injury, you will have to arrange for treatment on your own, as the study will not provide medical treatment or provide any compensation to you. You or your insurance provider will be billed for all costs of treatment for sickness or injury caused by the study. It is possible that your insurance will not cover these costs.

By signing this form, you do not give up your right to seek payment if you are harmed as a result of being in this study.

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

## 8.2 Will I be paid or given anything for taking part in this study?

No. You will not be paid for taking part in this study.

#### 8.3 Who could profit or financially benefit from the study results?

The company whose product is being studied: BMS

Information obtained from this study may help the University of Michigan learn more about the causes, risks, treatments, or how to prevent this and other health problems.

Research can lead to new discoveries, such as new tests, drugs, or devices. Researchers, their organizations, and other entities, including companies, may potentially benefit from the use of the data or discoveries. You will not have rights to these discoveries or any proceeds from them.

In the interest of transparency, we would like you to know that some of the researchers involved in this study have consulted for and/or held stock in BMS, may continue to do so, and may purchase or sell stock during the study period. These researchers are not likely to personally benefit from the results of this research.

## 9. CONFIDENTIALITY OF SUBJECT RECORDS AND AUTHORIZATION TO RELEASE YOUR PROTECTED HEALTH INFORMATION

The information below describes how the confidentiality of your research records will be protected in this study, and any sub-studies described in this document.

## 9.1 How will the researchers protect my information?

Your participation will occur at the University of Michigan medical center.

Your data will be kept confidential, to the extent permitted by applicable laws, in the following manner:

- Your name will not be used in any reports about the study
- You will be identified only by a study code: a patient ID number, and initials
- Your identifying information will be kept secure

The study team will assign a code number to the study data and may use your initials. Some study data may contain information that could be used (perhaps in combination with other information) to identify you (e.g., initials, date of birth).

The sponsor will use the study data for research purposes to support the scientific objectives of the study.

Study data (that does not directly identify you) may be published in medical journals or shared with others as part of scientific discussions.

## **Genetic Information Nondiscrimination Act (GINA)**

The federal Genetic Information Nondiscrimination Act (GINA) generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

your genetic information. This law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Under this law:

- Health insurance companies and group health plans may not request your genetic information that we obtain from this research
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums
- Employers with 15 or more employees may not use your genetic information that we obtain from this research when making a decision to hire, promote, or fire you or when setting the terms of your employment

GINA does not apply to the following groups, however these groups have policies in place that provide similar protections against discrimination:

- Members of the US Military receiving care through Tricare
- Veterans receiving care through the Veteran's Administration (VA)
- The Indian Health Service
- Federal employees receiving care through the Federal Employees Health Benefits Plans

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov/">http://www.clinicaltrials.gov/</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## 9.2 What protected health information (PHI) about me could be seen by the researchers or by other people? Why? Who might see it?

Signing this form gives the researchers your permission to obtain, use, and share information about you for this study, and is required in order for you to take part in the study.

Medical information and billing records are protected by the privacy regulations of the federal Health Insurance Portability and Accountability Act of 1996 (HIPAA). This type of information is called protected health information (PHI). PHI about you may be obtained from any hospital, doctor, and other health care provider involved in your care, including:

- Hospital/doctor's office records, including test results (X-rays, blood tests, urine tests, etc.)
- Mental health care records (except psychotherapy notes not kept with your medical records)
- Alcohol/substance abuse treatment records
- HIV/AIDS status
- Sexually transmitted disease and/or other communicable disease status
- Genetic counseling/genetic testing records
- Health plan/health insurance records
- All records relating to your condition, the study intervention you have received, and your response to the study intervention
- Billing information
- Demographic information
- Personal identifiers

IRBMED Informed Consent Template — 3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

There are many reasons why information about you may be used or seen by the researchers or others during or after this study. Examples include:

- The researchers may need the information to make sure you can take part in the study.
- The researchers may need the information to check your test results or look for side effects.
- University, Food and Drug Administration (FDA) and/or other government officials, auditors, and/or the IRB may need the information to make sure that the study is done in a safe and proper manner.
- Study sponsors or funders, or safety monitors or committees, may need the information to:
  - Make sure the study is done safely and properly
  - o Learn more about side effects
  - Analyze the results of the study
- Insurance companies or other organizations may need the information in order to pay your medical bills or other costs of your participation in the study.
- The researchers may need to use the information to create a databank of information about your condition or its study intervention.
- Information about your study participation may be included in your regular UMHS medical record
- If you receive any payments for taking part in this study, the University of Michigan accounting department may need your name, address, Social Security number, payment amount, and related information for tax reporting purposes.
- Federal or State law may require the study team to give information to government agencies. For example, to prevent harm to you or others, or for public health reasons.

The results of this study could be published in an article, but would not include any information that would let others know who you are.

## 9.3 What happens to information about me after the study is over or if I cancel my permission to use my PHI?

As a rule, the researchers will not continue to use or disclose information about you, but will keep it secure until it is destroyed. Sometimes, it may be necessary for information about you to continue to be used or disclosed, even after you have canceled your permission or the study is over.

Examples of reasons for this include:

- To avoid losing study results that have already included your information
- To provide limited information for research, education, or other activities. (This information would not include your name, social security number, or anything else that could let others know who you are.)
- To help University and government officials make sure that the study was conducted properly As long as your information is kept within the University of Michigan Health System, it is protected by the Health System's privacy policies. For more information about these policies, ask for a copy of the University of Michigan "Notice of Privacy Practices". This information is also available on the web at <a href="http://www.uofmhealth.org/patient+and+visitor+guide/hipaa">http://www.uofmhealth.org/patient+and+visitor+guide/hipaa</a>. Note that once your information has been shared with others as described under Question 9.2, it may no longer be protected by the privacy regulations of the federal Health Insurance Portability and Accountability Act of 1996 (HIPAA).

IRBMED Informed Consent Template — 3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

 Consent Subtitle: UMCC 2018.085
Consent Version: ICF v18Sep2020

## 9.4 When does my permission to use my PHI expire?

Your permission expires at the end of the study, unless you cancel it sooner. You may cancel your permission at any time by writing to the researchers listed in Section 10 "Contact Information" (below). If you withdraw your permission, you may no longer be eligible to participate in this study.

#### **10. CONTACT INFORMATION**

## 10.1 Who can I contact about this study?

Please contact the researchers listed below to:

- Obtain more information about the study
- Ask a question about the study procedures or treatments
- Talk about study-related costs to you or your health plan
- Report an illness, injury, or other problem (you may also need to tell your regular doctors)
- Leave the study before it is finished
- Express a concern about the study

Principal Investigator: Michelle Mierzwa, DM Mailing Address:

1500 E. Medical Center Drive

Ann Arbor, MI 48109

Telephone: (734) 845-3914

**Emergency Contact:** (734) 936-4000 (Hospital Operator – 24-hour paging)

## You may also express a question or concern about a study by contacting the Institutional Review **Board listed below:**

University of Michigan Medical School Institutional Review Board (IRBMED)

2800 Plymouth Road Building 520, Room 3214 Ann Arbor, MI 48109-2800

Telephone: 734-763-4768 (For International Studies, include the appropriate calling codes.)

Fax: 734-763-1234

e-mail: irbmed@umich.edu

If you are concerned about a possible violation of your privacy or concerned about a study you may contact the University of Michigan Health System Compliance Help Line at 1-866-990-0111. When you call or write about a concern, please provide as much information as possible, including the name of the researcher, the IRBMED number (at the top of this form), and details about the problem. This will help University officials to look into your concern. When reporting a concern, you do not have to give your name unless you want to.


Instructions revised 3-9-2018

DO NOT CHANGE THIS FIELD-IRB USE ONLY

#### 11. RECORD OF INFORMATION PROVIDED

## 11.1 What documents will be given to me?

Your signature in the next section means that you have received copies of all of the following documents:

• This "Consent to be Part of a Research Study" document. (Note: In addition to the copy you receive, copies of this document will be stored in a separate confidential research file and may be entered into your regular University of Michigan medical record.)


Other (specify):

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018

DO NOT CHANGE THIS FIELD—IRB USE ONLY

| 12. SIGNATURES |
|---|
| Consent/Assent to Participate in the Research Study |
| I understand the information printed on this form. I have discussed this study, its risks and potential benefits, and my other choices with |
| Print Legal Name: |
| Signature: |
| Date of Signature (mm/dd/yy): |
| Consent/Assent for Participating in an Optional Sub-Study: Blood Samples for Genetic Testing This project involves optional participation in a sub-study. I understand that it is my choice whether or not to take part in the sub-study. I understand that if my ability to consent or assent for myself changes, either I or my legal representative may be asked to re-consent prior to my continued participation in this study. |
| Yes, I agree to take part in the optional sub-study to collect blood samples for genetic testing. |
| No, I do not agree to take part in the optional sub-study to collect blood samples for genetic testing. |
| Print Legal Name: |
| Signature: |
| Date of Signature (mm/dd/yy): |

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018

 Consent Subtitle: UMCC 2018.085 Consent Version: ICF v18Sep2020

| Consent/Assent for use of Tumor Tissue Specimens for Unspecified Future Research This project involves the option to allow the study team to keep your identifiable specimens/data for use in future research. I understand that it is my choice whether or not to allow future use of my specimens. I understand that if my ability to consent or assent for myself changes, either I or my legal representative may be asked to re-consent prior to my continued participation in this study. |
|---|
| Yes, I agree to let the study team keep my specimens/data for future research. |
| No, I do not agree to let the study team keep my specimens/data for future research. |
| Print Legal Name: |
| Signature: |
| Date of Signature (mm/dd/yy): |
| Principal Investigator or Designee |
| I have provided this participant and/or his/her legally authorized representative(s) with information about this study that I believe to be accurate and complete. The participant and/or his/her legally authorized representative(s) indicated that he or she understands the nature of the study, including risks and benefits of participating. |
| Printed Legal Name: |
| Title: |
| Signature: |
| Date of Signature (mm/dd/yy): |

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018

DO NOT CHANGE THIS FIELD—IRB USE ONLY

UMCC 2018.085

"Latino."

## **PERSONAL CENSUS FORM**

| Na | me | | Date |
|---|---|---|---|
| Ce | e National Cancer Institute requires that The Un<br>inter report race and ethnicity information abou<br>ensure that all populations are offered the opp | ıt people | e who participate in clinical research |
| | Check here if you do not wish to provide some | or all of | the information below. |
| 1. | What race do you consider yourself to be? (Please select <i>one or more</i> ) | | American Indian/Alaska Native <sup>a</sup> Asian <sup>b</sup> Black or African American <sup>c</sup> Native Hawaiian or Other Pacific Islander <sup>d</sup> White <sup>e</sup> More than one race <sup>f</sup> |
| 2. | Do you consider yourself to be Hispanic <sup>g</sup> ? | ☐ Yes | no □ No |
| | merican Indian or Alaska Native- A person having origins uth America, and who maintains tribal affiliation or comn | | |
| suk | sian- A person having origins in any of the original people<br>ocontinent, including, for example, Cambodia, China, Indi<br>ands, Thailand and Vietnam. | | |
| | lack or African American- A person having origins in any cation and the same of the same o | | |
| | ative Hawaiian or Other Pacific Islander- A person having<br>moa, or other Pacific Islands. | origins in | any of the original peoples of Hawaii, Guam |
| e W | /hite- A person having origins in any of the original peopl | es of Euro | pe, the Middle East, or North Africa. |
| | lore than one race- (It is preferred that this be selected in ove, but this may also be solely selected.) | addition | to the selection of the specific races listed |
| | ispanic or Latino- A person of Mexican, Puerto Rican, Cub<br>ture or origin, regardless of race. The term "Spanish orig | | |